CLINICAL TRIAL: NCT06072547
Title: Effect of Flavored on!® Nicotine Pouch Products on Smoking Behaviors: a Sequential Multiple Assignment Randomized Controlled Trial
Brief Title: Effect of Flavored on!® Nicotine Pouch Products on Smoking Behaviors: a SMART Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Altria Client Services LLC (Industry)
Collaborators: Rose Research Center, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ALCS-REG-23-04-OTDN
Record Dates: First submitted 2023-09-29; First posted 2023-10-10 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Cigarette Smoking Behavior
Keywords: on! Nicotine Pouches; Reduction in Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Fruit; SPEN protein, human; Coffee

STUDY DESIGN:
Intervention Model Description: The study involves two randomizations, one at the beginning of the study and another at the end of week 3.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Complete flavor profile of on! nicotine pouches (Experimental): This study arm will provided with access to all varieties of 4mg on! nicotine pouch products throughout the trial.
  Interventions: Other: Access to all varieties of on! 4mg nicotine pouches (Berry, Citrus, Cinnamon, Wintergreen, Mint, Coffee, and Original)
- Non-Flavored on! nicotine pouches only (Active Comparator): This study arm will provided with access to non-flavored (i.e., Original) 4mg on! nicotine pouch products throughout the trial.
  Interventions: Other: Access to Original on! 4mg nicotine pouches
- Non-Flavored then complete flavor on! nicotine pouches (Active Comparator): This study arm will provided with access to non-flavored (i.e., Original) 4mg on! nicotine pouch products during the first 3 weeks of the trial and then access to all varieties of 4mg on! nicotine pouch products during the last 3 weeks of the trial.
  Interventions: Other: Non-Flavored then complete flavor on! nicotine pouches

INTERVENTIONS:
Other: Access to all varieties of on! 4mg nicotine pouches (Berry, Citrus, Cinnamon, Wintergreen, Mint, Coffee, and Original) — Access to all varieties of on! 4mg nicotine pouch products (Berry, Citrus, Cinnamon, Wintergreen, Mint, Coffee, and Original), throughout the trial.
  Other Names: Flavored on! nicotine pouches
  Arms: Complete flavor profile of on! nicotine pouches
Other: Access to Original on! 4mg nicotine pouches — Access to non-flavored (i.e., Original) 4mg on! nicotine pouch products throughout the trial.
  Arms: Non-Flavored on! nicotine pouches only
Other: Non-Flavored then complete flavor on! nicotine pouches — Access to non-flavored (i.e., Original) on! 4mg nicotine pouch products during the first 3 weeks and then access to all varieties (Berry, Citrus, Cinnamon, Wintergreen, Mint, Coffee, and Original) of on! 4mg nicotine pouch products during the rest of the trial
  Arms: Non-Flavored then complete flavor on! nicotine pouches

SUMMARY:
The goal of this clinical trial is to learn about the role of flavored on!® nicotine pouch products (the research products), an oral tobacco-leaf-free product, in the replacement of cigarettes with the use of the research products among adults who smoke cigarettes. The main question it aims to answer is whether flavored (vs. non-flavored) research products generate greater reduction of cigarette smoking among adults who smoke cigarettes.

Participants will be provided with research products to use for 6 weeks. Researchers will compare the reduction in cigarette smoking between participants with access to a complete flavor profile of research products and participants with access to only the Original (non-flavored) variety of research product to see if reduction in cigarette smoking is greater among those with access to flavored research products.

DETAILED DESCRIPTION:
This open label randomized controlled study (target n=400) among adults who smoke will evaluate the impact of differential availability of research products on cigarette smoking. All products will be on!® 4mg nicotine pouch products.

In this design, there are three configurations:

1. Access to complete flavor profile (Berry, Citrus, Cinnamon, Wintergreen, Mint, Coffee, and Original) for the entire six-week trial period (Group I);
2. Access to Original only for the entire six-week trial period (Group IIa); and
3. Access to Original only for the first three-week period and then access to complete flavor profile for the second three-week period (Group IIb).

This study will involve approximately 7 weeks (including the baseline period) of study participation in a home use test with daily surveys, weekly surveys, and a 6-month follow-up survey after the trial period. Approximately 400 participants will be recruited. A total of 150 participants will be randomized to Group I, 125 to Group IIa, and 125 to Group IIb.

After consenting and screening procedures, participants will be followed for 3-7 days to establish baseline measures of cigarettes smoked per day. During this baseline period at least two CO readings will be collected. Participants randomized into Group I will enter a seven-day trial period to try all flavors of research products. This trial period is intended to allow participants to identify their preferred flavor(s). After the trial period, they will then complete five additional weeks of home use testing with ad libitum product trial of research products with free choice of the flavors available in this study.

Likewise, following the baseline period, participants randomized into Group II will be provided with the Original variety of research products to use for the next three weeks. At the three-week point, participants in Group IIa will continue with the Original variety of research product for the remaining three weeks and Group IIb will switch to having access to all flavors of research products for the remaining three weeks. Group IIb will enter a seven-day trial period to try all flavors of research products (a total of seven packs - one of each flavor will be provided). This trial period is intended to allow participants to identify their preferred flavor(s). After the trial period, they will then complete two additional weeks of home use testing with ad libitum product trial of research products with free choice of the flavors available in this study.

Participants will be invited to complete a six-month follow-up survey to gain insights about their tobacco use and related factors after the end of the product trial.

Analysis will be conducted to compare outcomes between:

1. Group I vs. Group II at week 3
2. Group I vs. Group IIa at week 6
3. Group IIa vs. Group IIb at week 6 among non-responders at week3
4. Group IIa and Group IIb at week 6 among responders at week 3
5. Group I and Groups IIb at week 6

ELIGIBILITY:
Inclusion Criteria:

1. Has signed the Informed Consent Form (ICF) and is able to read and understand the information provided in the ICF.
2. Healthy adults who smoke cigarettes and are 22 to 65 years of age (inclusive) at screening.
3. Smokes an average of at least 5 cigarettes per day for the last 12 months.
4. Does not intend to use an FDA-approved treatment for nicotine dependence within the next 60 days (as assessed at screening).
5. Interested in replacing combustible cigarettes with a smoke-free tobacco product.
6. Willing and able to comply with the requirements of the study.
7. Owns a smart phone with text message and data capabilities compatible with necessary surveys.

Exclusion Criteria:

1. Participant enrollment numbers met (in sub-group or entire study).
2. Participant, or their first-degree relative (e.g., parent, sibling, child, spouse) or household member, is a current or former employee of the tobacco or e-vapor industry.
3. Participant, or their first-degree relative (e.g., parent, sibling, child, spouse) or household member is a named party or class representative in litigation involving a tobacco or e-vapor company.
4. Participant, or their first-degree relative (e.g., parent, sibling, child, spouse), or household member, is a current or former employee of a marketing consultant, market research firm, advertising or promotions agency, television or radio station, magazine or newspaper, government regulatory agency or public policy advocacy group, or law firm or legal department of a company.
5. Participant self-reports being "in poor health."
6. Participants of childbearing potential (CBP) who have a positive pregnancy test (as assessed at screening) or are nursing or planning to become pregnant during their participation.
7. Participant has an allergy/sensitivity to menthol or menthol-containing products or phenylalanine.
8. Participant has any other self-reported health restrictions.
9. Participant self-reports cardiovascular disease, cancer, diabetes, or is being treated for high blood pressure.
10. Participant self-reports periodontal disease, gum disease or bleeding, open mouth sores or ulcers.
11. Participant self-reports as wanting to stop using tobacco products in the next 60 days.
12. Participant has participated in one tobacco research study in the past 30 days OR a tobacco research study lasting two weeks or longer in the past 90 days.
13. Participant is unable to read, speak or understand English.
14. Participants who ever used at least a pack of nicotine pouch products or currently uses nicotine pouch products.
15. Participant who smokes marijuana more than once a week.
16. Heterosexually active participants of CBP (not sterilized by tubal ligation, oophorectomy, hysterectomy, or other surgical methods, or post-menopausal) that do not agree to practice medically appropriate methods of birth control (or remain abstinent) during the course of the trial and for 30 days after the last use of the research product. Medically acceptable methods of birth control include: vasectomy, vaginal diaphragm with spermicide, intrauterine device, hormonal birth control (oral, injected, patch, or implanted), condom with spermicide, or sponge with spermicide.
17. Taking psychoactive medications (e.g., antipsychotics or mood stabilizers).
18. Cannot participate in the study for any reason (e.g., medical, psychiatric, and or social reason) as judged by the Investigator or designated medical staff based on all available information from the screening period.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in cigarette-related toxicant exposure | End of Week 3, End of Week 6
  50% reduction in carbon monoxide (CO) readings from baseline (yes/no)
Cigarette-related toxicant exposure | End of Week 3, End of Week 6
  Reduction in numeric expired air CO readings

SECONDARY OUTCOMES:
Change in self-reported cigarette consumption | End of Week 3, End of Week 6
  50% reduction in self-reported cigarette consumption from baseline (Yes/No)
CO-verified smoking abstinence | End of Week 3, End of Week 6
  Cigarette smoking abstinence in the past 7 days based on self-report and CO<6ppm
Number of cigarettes smoked | End of Week 3, End of Week 6
  Numeric number of cigarettes smoked (based on self-report)

CONTACTS AND LOCATIONS:
Overall Officials: Hui Cheng, PhD, Principal Investigator — ALCS
Locations (1):
- Rose Research Center, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng HG, Rose JE, Karelitz JL, Botts DR, Botts TL, Willette PN, Cohen G. Effect of Flavored on! Nicotine Pouch Products on Smoking Behaviors: Protocol for a Sequential, Multiple Assignment, Randomized Controlled Trial. JMIR Res Protoc. 2024 Jun 21;13:e56565. doi: 10.2196/56565. PMID 38905632